CLINICAL TRIAL: NCT00128271
Title: A Phase 1 Study of Chimeric Anti-Phosphatidylserine Monoclonal Antibody (Bavituximab) in Patients Chronically Infected With Hepatitis C Virus (HCV) Who Are Non-Responders or Relapsers After Treatment With Pegylated Interferon Plus Ribavirin
Brief Title: Study of Bavituximab in Patients With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Dianne Uphoff/Senior Clinical Project Manager, Peregrine Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0501
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2006-08

CONDITIONS: Hepatitis C
Keywords: HCV; monoclonal antibody; phase 1
MeSH Terms: conditions — Hepatitis C | interventions — bavituximab

INTERVENTIONS:
Drug: Bavituximab

SUMMARY:
The purpose of this study is to determine the safety and tolerability of bavituximab when administered via a vein as a single infusion and to examine how bavituximab behaves in the body and how it affects the amount of hepatitis C virus in individuals with chronic infection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a world wide public health concern and is the most common chronic bloodborne infection in the United States and the leading indication for liver transplantation. Laboratory and animal studies have demonstrated that bavituximab binds viruses and virally infected cells and prolongs survival in infected animals. This study will examine the safety and tolerability of bavituximab when administered to patients with chronic HCV infection who do not respond to or relapse after treatment with pegylated interferon plus ribavirin combination therapy. Groups of patients will be treated with escalating doses and followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Chronic hepatitis C infection based on history and detectable serum HCV RNA
* Documented failure to respond to or relapse after treatment with pegylated interferon and ribavirin combination therapy
* Adequate hematologic function (absolute neutrophil count [ANC] greater than or equal to 1,500 cells/uL, hemoglobin [Hgb] greater than or equal to 12 g/dL in females and greater than or equal to 13 g/dL in males, platelet count greater than or equal to 100,000/uL and less than or equal to 500,000/uL)
* Adequate renal function (serum creatinine less than or equal to 1.5 mg/dL or calculated creatinine clearance greater than 60 mL/min)
* Normal coagulation profile (PT/INR and aPTT within institutional normal limits)
* D-dimer within institutional limits
* Female patients of childbearing potential must have a negative serum pregnancy test at prestudy and all patients of reproductive potential must be willing to use an approved form of barrier method contraception

Exclusion Criteria:

* Prior exposure to any chimeric antibody
* Any other cause of liver disease other than chronic hepatitis C, such as autoimmune or alcoholic liver disease
* Decompensated clinical liver disease or cirrhosis
* Any evidence of clinically significant bleeding
* Known history of bleeding diathesis or coagulopathy
* Any history of thromboembolic events including central venous catheter-related thrombosis
* Any evidence or history of a hypercoagulable state (eg, elevated d-dimer or shortened aPTT)
* Concurrent therapy with oral or parenteral anticoagulants
* Concurrent hormone therapy (ie, estrogen contraceptives, hormone replacement, anti-estrogen)
* Antiviral therapy within 90 days of day 0
* Investigational therapy within 4 weeks of day 0
* Major surgery within 4 weeks of day 0
* Uncontrolled intercurrent disease
* Any history of angina pectoris, coronary artery disease or cerebrovascular accident, or transient ischemic attack
* A history of any condition requiring anti-platelet therapy with the exception of general cardiovascular prophylaxis with aspirin
* A history of any condition requiring treatment (past or current) with coumarin-type agents
* Cardiac arrhythmia requiring medical therapy
* Serious non-healing wound
* Requirement for chronic daily treatment with NSAIDs, anti-platelet drugs (eg, phosphodiesterase inhibitors, adenosine diphosphate receptor antagonists), or steroids
* A disease or concurrent therapy known to cause significant alteration in immunologic function
* Known HIV or active hepatitis B virus (HBV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2005-08; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
adverse events
laboratory evaluations
human anti-chimeric antibody
pharmacokinetic analysis
viral kinetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Eliot W Godofsky, MD, FACP, Principal Investigator — Bach & Godofsky, MD, PA
Locations (1):
- Bach & Godofsky, MD, PA, Bradenton, Florida, United States